CLINICAL TRIAL: NCT06235099
Title: A Phase 3, Multi-Center, Open-label Study to Test the Diagnostic Performance of Copper Cu 64 PSMA I&T PET/CT in Men With Biochemical Recurrence of Prostate Cancer
Brief Title: Copper Cu 64 PSMA I&T PET Imaging in Men With Suspected Recurrence of Prostate Cancer
Acronym: Solar-Recur
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Curium US LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CURCu64PSM0002
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma; Biochemical Recurrence of Malignant Neoplasm of Prostate
Keywords: PSMA; Prostate Cancer; BCR; Solar-Recur; Cu-64 PSMA; PET; Solar
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic imaging with Copper Cu 64 PSMA I&T (Experimental): Copper Cu 64 PSMA I&T Injection
  Interventions: Drug: Copper Cu 64 PSMA I&T

INTERVENTIONS:
Drug: Copper Cu 64 PSMA I&T — Radiopharmaceutical PET imaging tracer injected intravenously for the detection of PSMA expression.

SUMMARY:
This is a prospective, open-label Phase 3 study to evaluate copper Cu 64 PSMA I&T injection for PET/CT imaging in patients with recurrent prostate cancer after radical prostatectomy or radiation therapy.

DETAILED DESCRIPTION:
The study will include approximately 200 patients with suspected biochemically recurrant prostate cancer. Each patient will be administered an 8 mCi (± 10 percent) intravenous dose of copper Cu 64 PSMA I&T injection. PET/CT imaging will be acquired for all patients at 1-4 hours ± 15 minutes post copper Cu 64 PSMA I&T injection.

The PET/CT images will be interpreted independently by three readers blinded to all patient information. Each patient study will be assessed and scored for the detection of prostate cancer. Specifically, each reader will categorize images as "Disease" or "No Disease" based only on tumor uptake of copper Cu 64 PSMA-I&T. Analysis of the reads will be used for determination of the patient-level correct detection rate and region-level correct localization rate of copper Cu 64 PSMA I&T PET/CT by comparison to the Reference Standard.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven prostate adenocarcinoma.
* Prior radical prostatectomy (greater than 6 weeks prior to screening) or radiation therapy (greater than 1 year prior to screening) with curative intent.
* Recurrence of disease defined as:

  1. Prior radical prostatectomy: PSA greater than or equal to 0.2 ng/mL followed by subsequent confirmatory PSA value greater than or equal to 0.2 ng/mL or
  2. Prior radiation therapy: 2 ng/mL rise in PSA over post-treatment nadir.
* Male aged greater than or equal to 18 years.
* Able to understand and provide signed written informed consent.

Exclusion Criteria:

* Androgen deprivation therapy (ADT) or other therapies targeting the androgen pathway within the past 3 months. Patients with a rising PSA level while on ADT for greater than 6 months are eligible.
* Patients participating in an interventional clinical trial within 30 days and having received an Investigational Product (IP) within five (5) biological half-lives prior to administration.
* Patients with any medical condition or circumstance (including receiving an IP or not capable of having a PET scan) that the investigator believes may compromise the data collected or lead to a failure to fulfill the study requirements.
* Patients who are planned to have an x-ray contrast within 24 hours or other PET radiotracer within 10 physical half-lives prior to the PET scan. If Barium contrast is administered this should be cleared before the PET scan.
* Patients who are administered any high-energy (greater than 300 keV) gamma-emitting radioisotopes within five (5) physical half-lives prior to copper Cu 64 PSMA I&T administration.
* Patients with known hypersensitivity to the active substance or any of the excipients of the IP.
* Patients who had a PSMA PET scan as part of their standard medical care within 90 days prior to enrollment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 235 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Patient-Level Correct Detection Rate (CDR) | 4 hours
  To determine the patient-level correct detection rate (CDR) of copper Cu 64 PSMA I&T injection PET/CT imaging for the detection of recurrent metastatic prostate cancer between 60 minutes to 240 minutes post injection. The CDR is defined as the percentage of patients who have at least one true PET positive lesion, with exactly localized correspondence between PET imaging and the Composite Reference Standard, regardless of any co-existent false positive findings, out of all patients who are scanned.
Region-Level Correct Localization Rate (CLR) | 4 hours
  To determine the region-level correct localization rate (CLR) of copper Cu 64 PSMA I&T injection PET/CT imaging for the detection of recurrent metastatic prostate cancer between 60 and 240 minutes post injection. The CLR is defined as the percentage of regions containing at least one true PET positive lesion, with exactly localized correspondence between PET/CT imaging and the Composite Reference Standard regardless of any co-existent false positive findings, within the same region, out of all regions containing at least one PET positive finding.

SECONDARY OUTCOMES:
CDR and CLR by Prostate-Specific Antigen level | 4 hours
  Comparison of patient level CDR and region level CLR of copper Cu 64 PSMA I&T PET/CT stratified by Prostate-Specific Antigen level.
CDR and CLR by histopathology available and histopathology unavailable | 4 hours
  Comparison of patient-level CDR and region level CLR of copper Cu 64 PSMA I&T PET/CT separated into subgroups of patients with histopathology available and unavailable.
Inter-reader and intra-reader agreement of copper Cu 64 PSMA I&T PET/CT interpretation on a per-patient basis | 4 hours
  Reader kappa statistics of copper Cu 64 PSMA I&T PET/CT scan interpretation by the blinded independent readers.
Incidence of adverse events of copper Cu 64 PSMA I&T injection | At time of dose administration up to 72 hours
  Treatment-emergent adverse events (AEs) will be assessed and graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Patient Level Detection Rate including subgroup analysis | 4 hours
  Endpoint elevated from exploratory to secondary.

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - Providence Medical Foundation, Fullerton, California
  - Tower Urology, Los Angeles, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - University of California, Irvine, Orange, California
  - San Francisco VA Medical Center, San Francisco, California
  - Providence Saint John's Health Center, Santa Monica, California
  - Stanford Hospital & Clinics, Stanford, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Miami Miller School of Medicine, Miami, Florida
  - Biogenix Molecular, LLC, Miami, Florida
  - Florida Urology Partners, Tampa, Florida
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Urology of Indiana, LLC, Carmel, Indiana
  - Indiana University Health Neuroscience Center, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - The University of Kansas Hospital, Kansas City, Kansas
  - M Health Fairview University of Minnesota Medical Center, Minneapolis, Minnesota
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - John Cochran VA Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Great Plains Health, Diagnostic Imaging, North Platte, Nebraska
  - XCancer, Omaha, Nebraska
  - Queens Hospital Center, Jamaica, New York
  - James J. Peters VA Medical Center, The Bronx, New York
  - Cleveland Clinic, Cleveland, Ohio
  - VA Portland Health Care System, Portland, Oregon
  - Carolina Urologic Research Center, LLC, Myrtle Beach, South Carolina
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Excel Diagnostics and Nuclear Oncology Center, Houston, Texas
  - Urology San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No